CLINICAL TRIAL: NCT02129491
Title: National Egyptian Network Pediatric Stroke and Hemiplegia Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics, Ain Shams University
Other Study IDs: NENPSHR
Record Dates: First submitted 2014-04-15; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Stroke With Hemiparesis; Perinatal Stroke; Focal Neurologic Deficits
Keywords: stroke; Congenital stroke; neonatal; hemiplegia
MeSH Terms: conditions — Neurologic Manifestations; Stroke; Hemiplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric Stroke and Hemiplegia: Any infant or child with acute stroke or hemiplegia

SUMMARY:
Our aim is to establish multi-center national Egyptian database of information about cerebrovascular stroke and hemiplegia in infants and children from 0 to 18 years of age.

DETAILED DESCRIPTION:
Aims: An open-ended multi-center, national Egyptian study to collect and analyze data for children with cerebrovascular stroke and hemiplegia .

Participants: Eligible infants and children with stroke and hemiplegia.

DESIGN: This study is a prospective cohort study.

Primary outcome measure: Initial acute stroke clinical and radiological presentation, recurrent stroke, mortality, and neurologic deficits in the acute stage, participants will be followed for the duration of hospital stay, an expected average of 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Focal neurological deficit of acute onset lasting greater than 20 minutes. And CT or MRI showing infarct in location consistent with neurological signs and symptoms
* Hemiplegia

Exclusion Criteria:

1. Cerebral haemorrhage not associated with ischemic infarct.
2. Hypoxic ischemic event with diffuse or bilateral infarction alone.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children from birth to 18 years of age with acute stroke presented by focal neurological signs confirmed by neuroradiology CT or MRI. All children with hemiplegia till the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Survival or neurologic deficit after acute cerebrovascular stroke. | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Children with acute stroke will be followed till either death or discharge from hospital, all clinical, radiological and therapeutic data will be collected.

SECONDARY OUTCOMES:
Long term neurological deficit | 12 months
  Post-stroke pediatric gross and fine motor function will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar MA Hassanein, MD, PhD, Study Chair — Pediatric Department, Children's Hospital, Faculty of Medicine, Ain Shams University
Locations (1):
- Pediatric Department, Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Abassia, Egypt

REFERENCES:
- See also: Faculty of Medicine, Ain Shams University — http://med.asu.edu.eg/
- See also: Ain Shams University web site — http://www.asu.edu.eg/